CLINICAL TRIAL: NCT01935076
Title: Placental miRNA (microRNA) Profile in Fetal Overgrowth Related to Maternal Obesity Study
Brief Title: miRNA in Fetal Overgrowth
Acronym: MIFO
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Celeste Durnwald, Assistant Professor, Maternal Fetal Medicine, Department of Obstetrics and Gynecology Director, Penn Perinatal Diabetes Program Director, High Risk Clinic at the Helen O. Dickens Center for Women's Health, University of Pennsylvania
Other Study IDs: 817124
Record Dates: First submitted 2013-08-19; First posted 2013-09-04 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: Maternal obesity; Macrosomic; miRNA; Fetal overgrowth
MeSH Terms: conditions — Obesity; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A small placental sample will be obtained after delivery in addition to cord blood collection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Obese mother/ Macrosomic baby: Obese mother that delivers a macrosomic neonate to understand the effects neonatal exposure to maternal obesity.
  Interventions: Behavioral: Neonatal exposure to maternal obesity
- Obese mother/ normal weight baby: Obese mother that delivers a normal weight neonate to understand effects neonatal exposure to maternal obesity.
  Interventions: Behavioral: Neonatal exposure to maternal obesity
- Normal weight mother/ Macrosomic baby: Normal weight mother that delivers a macrosomic neonate
- Normal weight mother/ Normal weight baby: Normal weight mother who delivered a normal weight neonate

INTERVENTIONS:
Behavioral: Neonatal exposure to maternal obesity
  Groups: Obese mother/ Macrosomic baby; Obese mother/ normal weight baby

SUMMARY:
The purpose of this study is to determine whether placental and umbilical cord blood miRNA expression is altered in women with obesity with macrosomic neonates to when compared to miRNA expression from control patients.

DETAILED DESCRIPTION:
MicroRNA's are a class of non-coding RNA's that function as translational repressors and are thought to modulate tissue development, proliferation, differentiation and function. Differential expression of certain placental miRNA's has been associated with preeclampsia.

The fetal origins of adult disease hypothesis suggests that risk factors from intrauterine environmental exposures affect the fetus' development during sensitive periods, and increases the risk of specific diseases in adult life. Our aim is to understand factors that predispose fetuses to fetal overgrowth in utero, especially in women with obesity. The objective of the study is to identify miRNA which are differentially expressed in the placenta and cord blood of pregnancies that are affected by fetal macrosomia to determine factors that may predispose fetuses to fetal overgrowth.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* prenatal care & delivery at the Hospital of the University of Pennsylvania system
* Normal glucose tolerance test results (less than 120 mg/dl)

Exclusion Criteria:

* Multiple gestation
* under 18 years old, or over 45 years old
* chronic hypertension
* preeclampsia
* chronic steroid use
* diabetes
* major fetal anomaly
* connective tissue disorder requiring medication
* active HIV
* Hepatitis C

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients delivering in the labor and delivery unit at the Hospital of the University of Pennsylvania.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Fetal Overgrowth | Delivery date to up to 6 weeks post partum
  Placental and cord blood samples will be studied for miRNA expression. The objective of the study is to identify miRNA which are differentially expressed in the placenta and cord blood of pregnancies that are affected by fetal macrosomia to determine factors that may predispose fetuses to fetal overgrowth.

CONTACTS AND LOCATIONS:
Overall Officials: Celeste P Durnwald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States